CLINICAL TRIAL: NCT06467994
Title: A Randomised, Controlled Trial Evaluating the Effectiveness of Boiled Cashew OraL immunoTherapy (BOLT) in Inducing Desensitisation or Remission in Children With Cashew Nut Allergy Compared With Placebo
Brief Title: Boiled Tree Nut for Oral Immunotherapy in Food-allergic Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Agnes Sze-Yin Leung, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOLT01
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Food Allergy in Children; Food Allergy
Keywords: food allergy; cashew allergy; tree nuts; oral immunotherapy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cashew Oral Immunotherapy (Active Comparator): Oral immunotherapy with boiled cashews followed by roasted cashews taken daily for 12 months
  Interventions: Other: Cashew oral immunotherapy
- Placebo Oral Immunotherapy (Placebo Comparator): Placebo oral immunotherapy taken daily for 12 months
  Interventions: Other: Placebo oral immunotherapy

INTERVENTIONS:
Other: Cashew oral immunotherapy — Cashew Flour (boiled/ roasted) that is prepared under food manufacturing regulations
  Arms: Cashew Oral Immunotherapy
Other: Placebo oral immunotherapy — Placebo oral immunotherapy consists of corn flour with food colouring that has similar appearance, taste and smell to the active product
  Arms: Placebo Oral Immunotherapy

SUMMARY:
As the global prevalence of food allergy steadily increases, tree nut (TN) becomes one of the main triggers of food-allergic reactions and food anaphylaxis. Since there is no effective cure, TN-allergic patients and their families must continue to live with this chronic, disabling condition while avoiding allergens and responding to allergic reactions with emergency treatment. An emerging experimental treatment for food allergy is oral immunotherapy (OIT). Tree nut OIT appears promising in preliminary studies but there are concerns about the high risk of adverse reactions to TNs used in the treatment. The rate of remission with TN OIT is also lacking. Identification of OIT regimes with increased efficacy and safety is urgently needed. The investigators revealed that boiled cashews had lower allergenic potential but retained mast cell reactivity. The aim of this proposed study is to investigate the efficacy and safety of a novel treatment strategy for TN-allergic individuals, whereby the investigators hypothesized that consuming increasing quantities of boiled cashews can induce desensitization/ remission to roasted tree nuts in children with cashew allergies.

DETAILED DESCRIPTION:
This will be a two-arm, parallel-design, double-blind, randomized controlled trial. Participants aged 3-17 years of age with double blind placebo-controlled food challenge-confirmed cashew allergy will be randomised into either the active or placebo arm. The active and placebo participants will consume daily dose of cashew and placebo, respectively, for 52 weeks. Participants will undergo an initial escalation and build-up phase until they reach a maintenance dose of cashew or placebo. Participants will return at 6 months for a safety and compliance check and at 12 months (T1) and 14 months (T2) for endpoint oral food challenges. Level of cross-desensitization to pistachio will be examined at T1. Immunological changes, including sIgE and IgG4, will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 3 year and 17 years of age;
* Either sex, and of any race and ethnicity;
* >7kg (the weight considered safe for the administration of an adrenaline autoinjector) (e.g. Jext);
* Confirmed diagnosis of cashew nut allergy as defined by a failed DBPCFC with cashew nut and a positive SPT (>=3mm than control) or sIgE to cashew nut (of at least 0.35 kUA) at screening.
* Subject's parent and/ or guardian must be able to understand and provide informed consent.

Exclusion Criteria:

* History of severe anaphylaxis (as defined by persistent hypotension, collapse, loss of consciousness, persistent hypoxia or ever needing more than three (3) doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Severe anaphylaxis during the study entry DBPCFC (defined as persistent hypotension, collapse, loss of consciousness, persistent hypoxia, or requiring more than 3 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Any disorder in which adrenaline is contraindicated (such as hypertension or cardiac rhythm disorders)
* Reacting to the placebo component during the study entry DBPCFC
* FEV1 <85% at rest and FEV1/FVC ≤ 85% at rest or ongoing chronic persistent asthma (as per Australian Asthma Foundation guidelines)
* Underlying medical conditions (e.g. cardiac disease) that increase the risks associated with anaphylaxis
* Use of beta-blockers, ACE inhibitors or calcium channel blockers
* Inflammatory intestinal conditions, indwelling catheters, gastrostomies, immune-compromised states, post-cardiac and/or gastrointestinal tract surgery, critically-ill and those requiring prolonged hospitalisation or other conditions that may increase the risks of probiotic associated sepsis
* Have received other food immunotherapy treatment in the preceding 6 months
* Currently taking immunomodulatory therapy (including allergen immunotherapy)
* Therapy with anti-IgE or other biologics within 1 year of enrolment
* Past or current major illness that in the opinion of the Site Investigator may affect the subject's ability to participate in the study e.g. increased risk to the participant
* History of suspected or biopsy-confirmed eosinophilic oesophagitis (EoE)
* Subjects who in the opinion of the Site Investigator are unable to follow the protocol NOTE: participants with other food allergies are NOT excluded from participating in this trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of cashew-allergic subjects who by T1 DBPCFC tolerate the full challenge i.e. a cumulative dose of 3180 mg cashew protein | T1 - One day after final day of maintenance treatment

SECONDARY OUTCOMES:
Proportion of participants with 8-week sustained unresponsiveness (passed T1 and T2 challenges) in OIT vs placebo groups | T2 - 8 weeks after final day of maintenance treatment
The cumulative dose tolerated during the T1 challenge (cumulative doses below the reaction-eliciting dose if there is a reaction; or total cumulative challenge dose if there is no reaction) in OIT vs placebo groups | T1 - One day after final day of maintenance treatment
Exposure-adjusted incidence rate and severity of treatment emergent adverse events (TEAEs) in OIT vs placebo groups; | T1 - One day after final day of maintenance treatment
SPT wheal size to cashew (at the end of treatment, and at 8 weeks after end of treatment) in OIT vs placebo groups. | T1 - One day after final day of maintenance treatment
Cashew-specific IgE levels (at the end of treatment, and at 8 weeks after end of treatment) in OIT vs placebo groups. | T1 - One day after final day of maintenance treatment
Cashew-specific IgG4 levels (at the end of treatment, and at 8 weeks after end of treatment) in OIT vs placebo groups. | T1 - One day after final day of maintenance treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- See also: Related Info — https://www.allergycuhk.org/bolt